CLINICAL TRIAL: NCT07151638
Title: Early Feasibility Trial for Fractomer™ Biomatrix: Safety Assessment in Healthy Human Participants
Brief Title: First-in-Human Safety Study for Fractomer™ Biomatrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: inSoma Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FRA-001
Record Dates: First submitted 2025-08-06; First posted 2025-09-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Soft Tissue; Soft Tissue Defects; Subcutaneous Injection
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Fractomer A (Experimental): Participants will be implanted with Fractomer A.
  Interventions: Device: Implantation (injection) of a new biomatrix for soft tissue support.
- Fractomer B (Experimental): Participants will be implanted with Fractomer B
  Interventions: Device: Implantation (injection) of a new biomatrix for soft tissue support.

INTERVENTIONS:
Device: Implantation (injection) of a new biomatrix for soft tissue support. — Implantation of a new injectable medical device, Fractomer Biomatrix, to study the safety of the product in healthy human participants.
  Other Names: Fractomer; implantable; bioresorbable medical device

SUMMARY:
The goal of this clinical trial is to evaluate the safety of implanting a new medical device (Fractomer™ Biomatrix) in healthy volunteers. The main question it aims to answer is:

How do healthy volunteers react to this injectable implant?

Participants will receive a subcutaneous injection of Fractomer and their health will be monitored. After the monitoring period, the implant will be removed.

DETAILED DESCRIPTION:
This clinical trial is designed to establish the safety of a new injectable device, which may provide a more effective means of treating deformations or voids in soft tissue. Healthy volunteers will be implanted in the subcutaneous space in the abdominal area, and health measures will be periodically recorded. The device will be removed per the protocol time periods, and the removed specimens will be examined for histological analysis by a trained pathologist. All data will be reviewed to determine the safety of this implanted, bioresorbable device.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 22 to 55.
4. Participants must be deemed by the Investigator to be generally healthy individuals based on a medical evaluation that includes a physical examination, medical history, vital signs, and the results from clinical, laboratory and other safety assessments collected during the Screening period. For medical history, there must be an absence of clinically significant diagnosis (in the opinion of the Investigator) of cardiovascular, dermatologic, endocrine, gastrointestinal, infectious, hematologic, hepatic, immunologic, metabolic, oncologic, neurologic, psychiatric, renal, or respiratory disease that may increase the risk of the participant in this study.

1. Participants with ongoing, stable anxiety and/or depression may be included, provided that they are stable and do not require the use of concomitant medications.

5. Ability to receive an injection of Fractomer™ and be willing to have a biopsy of the injection area be taken after either six weeks or three months.

6. For a person of child-bearing potential (POCBP)2: participant has a negative urine pregnancy test and has agreed to use contraceptives3 prior to and during their clinical trial participation.

7. BMI of 24 to 39.9, inclusive.

-

Exclusion Criteria:

* 1. Participant has, or the investigator believes them to have, a condition that would interfere with their ability to provide written informed consent, comply with study instructions, attend follow up visits, or which might confound the interpretation of the study results or put the subject at undue risk.

  2. Participants with any current or previous illness that, in the opinion of the investigator, might confound the results of the study or pose an additional, unacceptable risk to the participant or that could prevent, limit, or confound the protocol-specified assessments or study results' interpretation.

  3. Participant has or had a recent serious or ongoing infection, or risk for serious infection, or acute or chronic infection defined by the presence of any of the following:
  1. History of recurrent infections (defined as ≥ 3 infections requiring antimicrobial therapy within the 12 months prior to Screening).
  2. Hospitalization for infection or receipt of a course of intravenous (IV) antimicrobial therapy within 8 weeks prior to screening OR an opportunistic infection requiring hospitalization or IV antimicrobial treatment within 1 year of screening.
  3. Clinically significant chronic infection (e.g., osteomyelitis, bronchiectasis) within 8 weeks prior to Screening.
  4. Any herpes zoster, cytomegalovirus (CMV), or Epstein-Barr virus (EBV) infection that has not completely resolved within 12 weeks prior to Screening.
  5. History of splenectomy.
  6. Participant has hepatitis B or C virus or liver disease.
  7. Participant has a known seropositivity for, or active human immunodeficiency virus (HIV) infection.
  8. Participant is undergoing chemotherapy or has a history of malignancy
  9. Participant has collagen or elastin-vascular disease or other auto-immune disease.
  10. Participant is on immunosuppressive therapy.
  11. Or other condition(s) as indicated by the Investigator. 4. Participant has a history of type 1 or type 2 diabetes. 5. Participant has an allergy to lidocaine or epinephrine. 6. Participant has a hypersensitivity or allergy to adhesive tape. 7. Participant is pregnant or lactating. 8. Participant has a history of allergy or hypersensitivity to collagen or elastin injections.

      9. Participant is hypertensive (blood pressure 140/90 mmHg or higher), has cardiac or valvular disease, has a pacemaker or defibrillator, or has a known abdominal aortic aneurysm.

      10. Participant has blood coagulopathy. 11. Participant has a pre-existing skin condition, such as eczema, psoriasis, allergic dermatitis, scarring, or other condition, occurring bilaterally within the planned treatment area.

      12. Participant has a history of herpes in the planned treatment site. 13. Participant had radiation therapy or phototherapy, or current/active sunburn at the treatment site.

      14. Participant has a history of hyper- or hypo-pigmentation. 15. Participant has a history of keloid formation or poor wound healing. 16. Participant is concurrently enrolled in clinical trial at the time of screening, or has had exposure to any investigational agent, including topical agents, within 30 days or 5 half-lives prior to their enrollment visit, whichever is longer.

      17. Participant is an active, daily user of nicotine-containing products. 18. Participant is a user of recreational drugs as indicated by a positive result on drugs of abuse screen.
      1. If participant is user of THC products, participant may be included if they agree to stop use of THC products during their participation in this trial.
      2. If participant uses alcohol products, participant may be included if they limit their use to 2 or fewer alcohol units per day during their participation in this trial, and ingest no alcohol 48 hours before lab collection (site visit) timepoints.

      19. Participants who are intoxicated at time of enrollment.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2025-08-11 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with fever | Periodically over six weeks
  Each participant's temperature and signs of fever will be measured at each in-person visit as a measure of potential systemic reaction to the implanted device.
Number of participants with abnormal blood chemistry measures | Periodically over six weeks
  Participants will undergo blood draws at in-person visits to monitor serum chemistry. Any abnormal results that the investigator considers of concern will be flagged for follow-up. Each participant's blood chemistry will be measured at each in-person visit and evaluated as a measure of potential systemic reaction to the implanted device.
Number of participants with abnormal hematology results. | Periodically over six weeks
  Participants will undergo blood draws at in-person visits to monitor hematology/CBC profile. Any abnormal results that the investigator considers of concern will be flagged for follow-up. Each participant's CBC profile will be measured at each in-person visit and evaluated as a measure of potential systemic reaction to the implanted device.
Number of participants with abnormal coagulation results. | Periodically over six weeks
  Participants will undergo blood draws at in-person visits to monitor their coagulation profile. Any abnormal results that the investigator considers of concern will be flagged for follow-up. Each participant's coagulation profile will be measured at each in-person visit and evaluated as a measure of potential systemic reaction to the implanted device.
Number of participants with local signs of irritation or toxicity (observed at injection site) | Periodically over six weeks
  Participants will be examined at each in-person visit for any redness, swelling, bruising, pain, or tenderness at the injection site.
Number of participants with subjective signs of systemic response. | Periodically over six weeks
  Participants will undergo check-ins with investigators at in-person visits to monitor subjective signs of systemic reactions, including severe headaches or serious malaise. Any signs that the investigator considers of concern will be flagged for follow-up.
Number of participants with rejection or extrusion of the injection | Periodically over six weeks
  Participants will undergo check-ins with investigators at in-person visits to monitor the injection site, including an examination for any evidence of rejection or extrusion of the implanted device.
Number of SAEs | Periodically over six weeks
  Participants will undergo check-ins with investigators at in-person visits to monitor their health. Any SAE which is considered by the investigator to be injection- or device-related will be detailed and followed up per the protocol.

SECONDARY OUTCOMES:
Participant cellular responses to implanted device. | After the six week explant timepoint.
  Excised implants will be sent to expert pathologist assessment. The pathologist will note any observed peri-implant pathological response, including measures of inflammatory cell infiltrate, vascularization, fibrosis, notes on any residual implant, and the pathologist's overall conclusion on impact of the Fractomer™ implant.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Shamp, PhD, PA-C, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Saint Paul, Minnesota, United States